CLINICAL TRIAL: NCT04185480
Title: Evaluating Hemopatch in Reducing Seroma Related Complications Following Axillary Lymph Node Dissection: a Pilot Study
Acronym: HEIDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Principal Investigator, James van Bastelaar, Surgeon, Principal Investigator, MD, PhD, Zuyderland Medisch Centrum
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METCZ20190124
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Axillary Lymph Node Dissection; ALND; Axillary Clearance; Seroma
MeSH Terms: conditions — Seroma

STUDY DESIGN:
Intervention Model Description: A prospective cohort will be compared to a historical control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (No Intervention): Historical cohort of patients that underwent axillary clearance without hemopatch.
- Intervention (Experimental): Prospective cohort of patient undergoing axillary clearance with hemopatch
  Interventions: Device: Hemopatch

INTERVENTIONS:
Device: Hemopatch — Before closure of the wound this hemostatic sealant (Hemopatch), a pad of collagen derived from bovine dermis will be applied in the axilla
  Arms: Intervention

SUMMARY:
To evaluate if the use of Hemopatch in axillary lymph node dissection shows potential in reducing clinically significant seroma and seroma related complications, which might serve as a basis for a randomized controlled trial.

DETAILED DESCRIPTION:
Rationale:

Sentinel lymph node biopsy has reduced the number of patients needing to undergo axillary lymph node dissection (ALND). However, axillary lymph node dissection is part of curative therapy for a large group of patients with advanced invasive breast cancers and melanoma. Seroma may cause symptomatic discomfort requiring needle aspiration and is often associated with infection, wound dehiscence, skin necrosis, persistent fibrotic encapsulated seromas and may even delay adjuvant therapies [1]. Therefore, extensive research in finding the best technique in reducing seroma is needed.

Substances intended to seal small blood vessels by triggering collagen and fibrinogen synthesis supporting surgical hemostasis, are assumed to be able to contribute to sealing of these lymphatic vessels. Contradicting results were found in the effect of several fibrin-glue coated collagen patches [2-5] and fibrin glue [6,7]. Furthermore, the use of electrothermal bipolar vessel sealing system (LigaSure) in axillary dissection showed no significant reduction in rate of aspiration of seroma [8].

This pilot study is intended to assess the value of a haemostatic sealant (Hemopatch), a pad of collagen derived from bovine dermis, coated with NHS-PEG (pentaerythritol polyethylene glycol ether tetra-succinimidyl glutarate), in reducing seroma related complications after ALND with the advantage that this sealant is pliable and flexible.

Objective:

To evaluate if the use of Hemopatch in axillary lymph node dissection shows potential in reducing clinically significant seroma and seroma related complications, which might serve as a basis for a randomized controlled trial.

Study design:

A prospective cohort will be compared to a historical control group. Eighteen consecutive patients will undergo axillary lymph node dissection and after completion of lymphadenectomy, Hemopatch will be applied to the axillary surgical field. These results will be compared to the results of a historical control group consisting of 46 patients who have undergone ALND without the Hemopatch between January 2014 and December 2018.

Follow-up will be conducted for three months postoperatively.

Study population:

Patients of 18 years or older, diagnosed with stage III melanoma or breast cancer and indication for wide local excision (WLE) and/or axillary lymphadenectomy (ALND).

Intervention (if applicable):

Application of Hemopatch after standard axillary lymph node dissection.

Main study parameters/endpoints:

Proportion of patients treated with Hemopatch who develop clinically significant seroma.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Patients will be informed about the study before inclusion in the outpatient clinic. Informed consent will be obtained in the outpatient clinic a week after patients were initially informed. Postoperative check-ups will be done more frequently. Standard postoperative check-ups are planned at one week and three months. Additional study postoperative check-up will be performed at six weeks. Therefore, patients will be required to undergo one additional check-up. During out patients' visits, the wound will be evaluated and patients will be asked to fill in a questionnaire. Application of the Hemopatch is expected to reduce clinically significant seroma after ALND. The only potential risk for the patient is that the Hemopatch is ineffective.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of 18 years or older.
* Patients with melanoma and indication for axillary lymph node dissection.
* Patients with breast cancer and indication for breast conserving therapy and axillary lymph node dissection
* Patients with an indication for secondary axillary lymph node dissection.

Exclusion Criteria:

* Patients with breast cancer who have an indication for modified radical mastectomy.
* Unable to comprehend implications and extent of study and sign for informed consent
* Pregnant women
* Patients included in another breast related clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients treated with Hemopatch who develop clinically significant seroma during the first three post-operative months | During the first three postoperative months
  Proportion of patients treated with Hemopatch who develop clinically significant seroma during the first three post-operative months. Clinically significant seroma defined as:
  1. Wound healing is at risk due to seroma (wound break down, seroma leakage, necrosis) and possibly operative debriding of the wound or use of vacuum assisted wound therapy is necessary.
  2. The presence of discomfort or pain caused by large amounts of seroma, characterised by tenseness of the skin and aspiration is necessary
  3. The presence of contaminated/ infected seroma, and aspiration is necessary to treat infection. All patients that undergo seroma aspiration due to infection will also be treated with a one week course of Augmentin 625 mg 3 times daily.
  4. Seroma for which incision and drainage is necessary to treat abscess or infection.

SECONDARY OUTCOMES:
Surgical site infection (SSI) rate | During the first three postoperative months
  Surgical site infection (SSI) rate, defined as redness, pain, heat or swelling at the site of the incision or by the drainage of pus. Infection rate will be measured by A) the need for antibiotics, B) seroma aspiration due to infection or C) surgical drainage during the first three postoperative months.
The number of outpatient department visits | During the first three postoperative months
  Number of unplanned visits to the ER or outpatient clinic. Planned visits are standard follow-up outpatient clinic visits which are defined preoperatively. Unplanned visits are defined as any visit to the outpatient clinic which is necessary due to an adverse event.
Number of days before removal of axillary drainage and axillary drainage output. | During the first three postoperative months
  Number of days before removal of axillary drainage and axillary drainage output. According to current guidelines the drain is always removed no later than five days, earlier if drain output is < 50 ml/ 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Zuyderland Medisch Centrum, Sittard, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No